CLINICAL TRIAL: NCT06497920
Title: Modulating Plasticity in the Motor Cortex Using Repetitive Transcranial Magnetic Stimulation to Improve Motor Function in Autism Spectrum Disorder
Brief Title: rTMS to Improve Motor Function in Autism
Acronym: (AMBLE Autism)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023/180
Record Dates: First submitted 2024-06-13; First posted 2024-07-12 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder; Motor Activity
Keywords: Autism; Motor Function; Repetitive Transcranial Magnetic Stimulation; Transcranial Magnetic Stimulation; Motor Cortex; Electroencephalography
MeSH Terms: conditions — Autism Spectrum Disorder; Motor Activity; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: This project includes a randomized controlled trial. We will use a randomized, double- blind, sham-controlled design comparing the efficacy of active vs. sham rTMS (6000 pulses at 20 Hz/session, 3000 pulses/hemisphere with 5-10 min break in between) delivered to the motor cortex using bilaterally, 1 session/day for 3 consecutive days (3 sessions). Pulses will be delivered to one hemisphere (left or right) first, followed by the opposite side. The sequence will be randomized for each participant.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent assistant external to the project will manage the randomization of subjects. The clinician, investigators, participant and technician will all be blinded. To ensure blinding during treatment, either the active or sham adapter will be connected to the Magstim Horizon, the coil will remain the same. To ensure blinding of the technician and the participant an independent study assistant will connect the active or sham adapter for the Magstim Horizon. Both heads have identical external appearances, and stimulation of either coil generates identical auditory and somatosensory (vibration) stimuli. All raters obtaining outcome measures will also be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS (Active Comparator): Autistic adults receiving active rTMS to the motor cortex.
  Interventions: Device: Active rTMS to the motor cortex
- Sham rTMS (Sham Comparator): Autistic adults receiving sham rTMS to the motor cortex.
  Interventions: Device: Sham rTMS to the motor cortex

INTERVENTIONS:
Device: Active rTMS to the motor cortex — Active bilateral repetitive transcranial magnetic stimulation to the motor cortex
  Arms: Active rTMS
Device: Sham rTMS to the motor cortex — Sham bilateral repetitive transcranial magnetic stimulation to the motor cortex
  Arms: Sham rTMS

SUMMARY:
In the current project, investigators have two main goals: i) Testing whether an excessive plasticity, i.e. hyperplasticity in the motor cortex underlies motor function difficulties in autistic adults, and ii) Using repetitive Transcranial Magnetic Stimulation (rTMS) with autistic adults to examine whether resulting reduced hyperplasticity in the motor cortex will be associated with clinical improvements in the motor function.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a very common developmental condition, yet the cause remains unknown and effective treatment options to improve outcomes remain limited. Most autistic adults experience significant motor function difficulties involving balance, posture, coordination, and strength that negatively affect their quality of life, social interaction, confidence and daily functioning. Therefore, such difficulties remain an important treatment target. However, there are no known effective clinical interventions for such difficulties. Investigators previously showed that the part of the brain that controls motor movements, i.e. motor cortex, showed hyperplasticity, as assessed by theta-burst magnetic brain stimulation (TBS), in autistic adults. Hyperplasticity may adversely affect brain health and behavior. Investigators also previously found that rTMS may reduce such hyperplasticity in the motor cortex in autistic adults.

In this project, 100 autistic adults with significant motor function difficulties and 50 neurotypical (NT) controls matched 2:1 based on age, sex, and IQ will be recruited. At the Centre for Addiction and Mental Health, Toronto, each autistic adult's participation will consist of eight visits, while each NT adult's participation will include two visits.

All participants, both autistic and NT, will undergo clinical, adaptive, and motor function assessments during their first visit (lasting approximately 3 hours) and a pre- and post-intermittent-TBS (iTBS) session, paired with electroencephalography (EEG), to induce and assess plasticity in the left or right motor cortex (depending on handedness) during their second visit (lasting approximately 3 hours). Based on the preliminary evidence that rTMS reduces hyperplasticity in the motor cortex in autistic adults, the investigators will then use a randomized, double-blind, sham-controlled design for bilateral 3-session rTMS on the motor cortex. Autistic participants will be randomized (1:1, sex-stratified) to receive either active or sham rTMS (150 trains of 40 pulses with an inter-train interval of 25 seconds, delivered at 90% of the resting motor threshold for both conditions) three days a week (approximately 1.5 hours each), from their third to fifth visits (total of 3 sessions). Assessment of motor and adaptive function, and plasticity in the motor cortex will be repeated the next day, one week (seventh visit), and four weeks (eighth visit) after the last rTMS session (i.e. 3rd rTMS session).

ELIGIBILITY:
Inclusion Criteria:

ASD or control participants must meet all of the inclusion criteria to eligible for this study:

1. Aged between 18 and 40 years old. 40 years is chosen as the cut-off because of the report of high rates of Parkinsonism in autistic adults > 39years;
2. Have IQ>70;
3. Are able to read, write and communicate effectively in English;
4. Are able to provide informed consent. We will recruit only intellectually-able autistic adults. The intellectual ability will be determined using WASI-II. The ability to provide consent will be determined using clinical assessment.
5. Have no prior history of seizure;
6. Must sign and date the informed consent form;
7. Stated willingness to comply with all study procedures;
8. Agreement to adhere to Lifestyle Considerations, that is: refrain from consumption of alcohol, tobacco, marijuana, or caffeine on the day of study visits.

All ASD participants:

1. Will have DSM-5 diagnosis of ASD without intellectual disability, confirmed by clinical assessment and the Autism Diagnostic Observation Schedule - 2 (ADOS-2);
2. Will have significant motor function difficulties defined as a standard composite score <40 (i.e., >1 standard deviation below the mean) on either fine or gross motor composite scores of the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition or BOT-2;
3. Are clinically stable as determined by clinical assessment, with no medication changes over the past 4 weeks. Given the high variability of handedness in ASD, we will include participants with left, right or mixed handedness.

Exclusion Criteria:

ASD or control participants will be excluded if they experience/have:

1. Current pregnancy;
2. Current or past history of co-morbid medical condition that may require urgent medical intervention;
3. DSM-5 substance use disorder (other than tobacco) within the past 6 months; however, all participants will be asked to refrain from smoking or taking caffeine four hours prior to the iTBS session;
4. Significant hearing or visual impairment interfering with the ability to read or hear instructions;
5. Significantly debilitating medical or neurologic illness (e.g., encephalitis, aneurysms, tumors, central nervous system infections), or acute or unstable medical illnesses as determined by project physician (e.g., uncontrolled diabetes);
6. Metal implants or a pace-maker;
7. Prior rTMS treatment;

In addition, ASD participants will be excluded if they report taking benzodiazepines or anticonvulsants currently.

NT controls will be excluded if they have:

1. Presence of psychopathology other than specific phobia, as screened by Personality Assessment Inventory and;
2. A known diagnosis of Pervasive Developmental Disorder or ASD among any biologically related family members.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in motor cortical plasticity using motor evoked potentials (MEPs) in autistic adults following rTMS. | Plasticity in the motor cortex will be evaluated at baseline, the day after the final rTMS session, and again at 1 and 4 weeks after the last rTMS session.
  Plasticity will be indexed by the duration of facilitation of motor evoked potentials (MEPs) amplitude, i.e. the time for the MEP amplitude to return to baseline values following iTBS.
Changes in motor function in autistic adults following rTMS. | Motor function will be assessed at baseline, the day after the final rTMS, and again at 1 and 4 weeks after the last rTMS session.
  Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) will be used to assess motor function. The total motor composite score will be used as the primary measure of motor function. A higher score on BOT-2 indicates better motor performance.

SECONDARY OUTCOMES:
Changes in motor cortical plasticity using cortical evoked activity (CEA) in autistic adults following rTMS. | Plasticity in the motor cortex will be evaluated at baseline, the day after the final rTMS, and again at 1 and 4 weeks after the last rTMS session.
  A secondary measure of plasticity will be indexed by the maximum post-iTBS/pre-iTBS cortical evoked activity (CEA) ratio. CEA will be defined as the area under rectified curve for averaged electroencephalography (EEG) recordings in the electrode over motor cortex between 50-275 millisecond post-stimulus.
Changes in the adaptive daily living skills in autistic adults following rTMS. | Adaptive daily living skills will be assessed at baseline, the day after the final rTMS, and again at 1 and 4 weeks after the last rTMS session.
  The daily living skills domain of Adaptive Behavior Assessment System-3rd edition will be used to assess adaptive daily living skills. A higher score represents better adaptive skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Addiction and Mental Health (CAMH), Toronto, Ontario, Canada

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT06497920/Prot_SAP_000.pdf